CLINICAL TRIAL: NCT06820177
Title: Prophylactic Tranexamic Acid for Second Trimester Dilation and Evacuation and Bleeding Outcomes: A Randomized Controlled Trial
Brief Title: Tranexamic Acid for Second Trimester Dilation and Evacuation and Bleeding Outcomes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sarah Averbach, MD MAS, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 811490
Record Dates: First submitted 2025-02-04; First posted 2025-02-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-02

CONDITIONS: Abortion; Dilation and Evacuation; Hemorrhage; Prophylactic Tranexamic Acid Use; Blood Loss
Keywords: abortion; dilation and evacuation; TXA; hemorrhage; Tranexamic acid; D&E
MeSH Terms: conditions — Dilatation, Pathologic; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 10 mL of normal saline administered via IV at the start of the D&E procedure
  Interventions: Drug: Placebo
- Tranexamic acid (Active Comparator): 1g tranexamic acid administered via IV at the start of the D&E procedure
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 1g tranexamic acid
  Arms: Tranexamic acid
Drug: Placebo — 10 mL 0.9% normal saline
  Arms: Placebo

SUMMARY:
Although procedural abortion in the second trimester is extremely safe, hemorrhage is one of the leading causes of morbidity and mortality. Tranexamic acid (TXA) is used commonly in obstetrics to prevent or manage intrapartum or postpartum hemorrhage and has been associated with decreased mortality and decreased blood loss at the time of birth. Some guidelines are recommending the use of TXA for both the prevention and management of bleeding for abortion care. However, there are currently no published studies assessing the association between TXA and bleeding outcomes for abortion procedures. This study will involve a randomized, placebo-controlled trial of pregnant patients aged 18 and older desiring dilation and evacuation (D&E) for abortion or fetal demise at 18-24 weeks gestation. The primary aim is to determine whether prophylactic TXA has an effect on the need for additional interventions to control bleeding at the time of D&E. The secondary aim is to determine whether prophylactic TXA has an effect on the mean quantitative procedural blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign informed consent
* Speaks English or Spanish language,
* Requesting pregnancy termination or procedural management of fetal demise - Intrauterine pregnancy, 18 weeks 0 days and 24 weeks and 0 days gestation

Exclusion Criteria:

* History of or current thromboembolic event (deep vein thrombosis, stroke, pulmonary embolism)
* History of coagulopathy
* Anticoagulant use in the preceding five days
* Severe renal impairment
* Chorioamnionitis or sepsis
* Suspected placenta accreta spectrum
* Prophylactic uterotonics other than oxytocin given (or planned to be given) at the start of the D&E
* Known allergic reaction or hypersensitivity to TXA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of excessive bleeding | During the D&E procedure or immediately after
  The use of any of the following interventions to manage excessive bleeding: at least one uterotonic medication given (i.e. methylergonovine maleate, carboprost tromethamine, misoprostol or additional oxytocin after the standard 30 units), blood transfusion, re-aspiration for bleeding or hematometra, intra-uterine balloon tamponade, uterine artery embolization, major surgery for bleeding, admission for bleeding, or prescription given for any uterotonic medication at discharge.

SECONDARY OUTCOMES:
Mean intra-operative quantitative blood loss | During the D&E procedure
  Blood loss measured from the start of the procedure (after removal of cervical dilators) until the end of the procedure (after removal of the speculum). Blood loss will be measured in mL by collecting the blood in a draped bag underneath the patient and weighing all gauze/chux used during the procedure.
Mean post-operative quantitative blood loss | on the day of the procedure up to 4 hours following the procedure
  Any bleeding that occurs after speculum removal in the procedural room until the patient leaves clinic on the day of the procedure up to 4 hours following the procedure. The patient's menstrual pad(s) in the recovery room will be weighed.
Total number of interventions to control bleeding | During the D&E procedure or immediately after
  The total number of interventions performed within the primary composite outcome will be assessed.
Individual interventions used to control bleeding for each participant | During the D&E procedure or immediately after
  Individual outcomes within the primary composite outcome will be assessed.
Number of doses of uterotonics given | During the D&E procedure or immediately after
  We will assess the number of doses of uterotonics given for each participant
Provider satisfaction with bleeding outcomes | Immediately after the D&E procedure
  Each D&E provider will be asked about their satisfaction with bleeding outcomes for the procedure using a 5 point Likert scale (from 0 being very unsatisfied to 5 being very satisfied).
Provider assessment of which treatment assignment they believe the participant received | Immediately after the D&E procedure
  D&E providers will be asked if they think the participant received the study drug or placebo.
Length of the procedure | During the D&E procedure
  The length of the D&E procedure will be recorded in minutes from the time the speculum is first instrument is placed in the uterus until the speculum is removed (minus any time for IUD placement).
Adverse events | During the D&E procedure or immediately after
  Adverse events will be assessed including: thromboembolic event, nausea, vomiting, dizziness or hypersensitivity will be ascertained on day of the procedure and by patient self report after

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - Planned Parenthood of the Pacific Southwest, San Diego, California

IPD SHARING:
Plan to Share IPD: No